CLINICAL TRIAL: NCT00004467
Title: Randomized Study of Acetylcysteine in Patients With Acute Liver Failure Not Caused by Acetaminophen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 199/13925 DK52827 (completed); R03DK052827 (NIH); UTSMC-IRB-0697-27200 (Other: University of Texas Southwest Medical Center); R01DK058369 (NIH); U01DK058369 (NIH); NCT00587366 (obsolete NCT alias)
Expanded Access: Available
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Acute Liver Failure
Keywords: acute liver failure; gastrointestinal disorders; rare disease
MeSH Terms: conditions — Liver Failure, Acute; Gastrointestinal Diseases; Rare Diseases | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- N-acetylcysteine (NAC) (Experimental)
  Interventions: Drug: N-acetylcysteine (NAC)

INTERVENTIONS:
Drug: N-acetylcysteine (NAC) — Infusion of 5% dextrose with N-acetylcysteine with an initial loading dose of 150 mg/kg/h of NAC over 1 hour, followed by 12.5 mg/kg/h for 4 hours, then continuous infusions of 6.25 mg/kg/h for the remaining 67 hours.
  Other Names: Acetadote
  Arms: N-acetylcysteine (NAC)
Drug: Placebo — Infusion of 5% dextrose
  Arms: Placebo

SUMMARY:
OBJECTIVES:

I. Determine the safety and efficacy of a short course (72 hours) of intravenous acetylcysteine in patients with acute liver failure for whom no antidote or specific treatment is available.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, multicenter study. Patients are randomized to receive intravenous acetylcysteine or placebo for 72 hours. Treatment must begin within 12 hours of hospitalization. Patients who advance to grade III or IV encephalopathy are eligible for liver transplantation.

Patients are followed at 3 weeks.

ELIGIBILITY:
Inclusion Criteria

This is a phase III blinded study, which will involve approximately 200 patients. For this purpose, acute liver failure will be defined as onset of any mental status alteration and coagulopathy (INR > 1.5) within 26 weeks of onset of a hepatitic illness, with no evidence of underlying chronic liver disease. Eligible patients will be those admitted to study site hospital intensive care units with acute liver failure and who can be evaluated and started on treatment within the first 24 hours of hospitalization or those who evolve to altered mentation if already in the hospital. All subjects will be between 18 and 70 years. Patients transferred from referring hospitals to a study site may be considered for enrollment, provided that no other specific treatment protocol has begun, and that no liver support device (bioartificial liver (BAL), extracorporeal liver assist device (ELAD), transgenic pig perfusion) has been used or is contemplated. Use of fresh frozen plasma infusions will not disqualify patients from participation.

Exclusion Criteria

1. Patients less than age 18 or over 70 years of age.
2. ALF patients where acetaminophen or mushroom poisoning is assessed or Suspected to be a significant contributing or sole cause of the illness. Both these diagnoses require specific antidote therapy, including NAC in the case of acetaminophen, rather than randomized or non-specific treatment.
3. Patients with a diagnosis of shock liver (ischemic hepatopathy), since the overall outcome for these patients in largely determined by the underlying etiology of the condition leading to shock. Heat stroke is not excluded.
4. Acute liver failure of pregnancy or the HELLP syndrome (pregnancy associated hemolysis and coagulopathy). The effect of NAC on the fetus or the mother has not been determined; in addition, pregnancy-related liver diseases usually mandate rapid delivery of the infant.
5. ALF thought secondary to intrahepatic malignancy. Patients with hepatic malignancy experiencing ALF have 100% mortality and are not transplant candidates.
6. Patients who exhibit signs of cerebral herniation at the time of enrollment.
7. Patients who demonstrate the presence of intractable arterial hypotension (arterial systolic blood pressure equal to or below 70 mmHg) present, or require inotropic drugs at the time of enrollment.
8. Severe sepsis (temperature >39o C and/or significant bacteremia) present at the time of enrollment.

In general, acute liver failure (ALF) patients comprise somewhat more women than men, but there is no preponderance of any racial group, other than that expected on the basis of geographic differences. No exclusion will be made on the basis of race, ethnic group or gender. Criteria for inclusion of women and minorities will be those established in the NIH guidelines. Each study site will provide for review a log of patients considered for the NAC study with no identifiers, yielding only gender and age, race and reason for not participating as a check on gender or ethnic bias.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 1998-06; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | 3 weeks

SECONDARY OUTCOMES:
Survival without liver transplantation (Spontaneous Survival | 3 weeks
Transplant rate | 3 weeks
Length of hospital stay | 3 weeks
Number of organ systems showing failure | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William M. Lee, MD, Study Chair — University of Texas Southwestern Medical Center at Dallas, Dallas, TX
Locations (25):
- United States (25):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - University of California Los Angeles, Los Angeles, California
  - University of California Davis, Sacramento, California
  - University of California San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Mayo Clinic, Jacksonville, Florida
  - Northwestern University Medical School, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai Medical Center, NY, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Result] Lee WM, Hynan LS, Rossaro L, Fontana RJ, Stravitz RT, Larson AM, Davern TJ 2nd, Murray NG, McCashland T, Reisch JS, Robuck PR; Acute Liver Failure Study Group. Intravenous N-acetylcysteine improves transplant-free survival in early stage non-acetaminophen acute liver failure. Gastroenterology. 2009 Sep;137(3):856-64, 864.e1. doi: 10.1053/j.gastro.2009.06.006. Epub 2009 Jun 12. PMID 19524577
- [Derived] Stravitz RT, Fontana RJ, Karvellas C, Durkalski V, McGuire B, Rule JA, Tujios S, Lee WM; Acute Liver Failure Study Group. Future directions in acute liver failure. Hepatology. 2023 Oct 1;78(4):1266-1289. doi: 10.1097/HEP.0000000000000458. Epub 2023 May 16. PMID 37183883
- [Derived] Singh S, Hynan LS, Rule JA, Lee WM. Changes in alpha-foetoprotein and Gc-globulin in relation to outcomes in non-acetaminophen acute liver failure. Liver Int. 2019 Dec;39(12):2368-2373. doi: 10.1111/liv.14216. Epub 2019 Sep 10. PMID 31421008
- See also: Acute Liver Failure Study Group — http://www.acuteliverfailure.org